CLINICAL TRIAL: NCT00992472
Title: Bioavailability of Prochlorperazine Suppositories, 25 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1670110293
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Healthy

ARMS (2):
- Prochlorperazine suppositories, 25mg (Experimental)
  Interventions: Drug: Prochlorperazine suppositories, 25mg
- Compazine® suppositories, 25mg (Active Comparator)
  Interventions: Drug: Compazine® suppositories, 25mg

INTERVENTIONS:
Drug: Prochlorperazine suppositories, 25mg
  Arms: Prochlorperazine suppositories, 25mg
Drug: Compazine® suppositories, 25mg
  Arms: Compazine® suppositories, 25mg

SUMMARY:
The purpose of this study is to compare prochlorperazine plasma concentrations produced after administration of the test formulation with those produced after administration of a marketed reference product.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by lack of clinically significant abnormalities in health assessment performed at screening

Exclusion Criteria:

* Positive test results for HIV or Hepatitis B or C
* History of allergy or sensitivity to Prochlorperazine or related drugs

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Ferguson, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.
Locations (1):
- PharmaKinetics Laboratories, Inc, Baltimore, Maryland, United States